CLINICAL TRIAL: NCT04645758
Title: The Immediate Effects of Dry Needling and Extra Corporeal Shockwave Therapy on Hand Grip Strength.A Randomised Controlled Trail.
Brief Title: A Study to Analyse the Immediate Effect of Dry Needling and Extra Corporeal Shock Wave Therapy on Hand Grip Strength
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Comprehensive Rehabilitation Centre, Medina, Saudi Arabia (Other)
Responsible Party: Principal Investigator, Rayan Mohammed Al Fadani, Head of the Department of Physical therapy and Rehabilitation., Comprehensive Rehabilitation Centre, Medina, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Rct001
Record Dates: First submitted 2020-09-22; First posted 2020-11-27 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Muscle Weakness Condition
Keywords: Dry needling; Extra corporeal Shockwave therapy; Hand Grip Strength; Post 1 hour
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: M.M.K outcome blind assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling Group or (DN) (Active Comparator): Dry needling for 5 mins on the flexor group of muscles of dominant forearm.
  Interventions: Combination Product: Dry needling and Extra corporeal Shock wave therapy
- Extra corporeal Shockwave therapy Group or (ESWT) (Active Comparator): Delivering of Shock wave pulses of 1250 at the energy intensity of 0.58 mj/mm2 on the flexor group of muscles of dominant forearm
  Interventions: Combination Product: Dry needling and Extra corporeal Shock wave therapy

INTERVENTIONS:
Combination Product: Dry needling and Extra corporeal Shock wave therapy — 5 mins of dry needling and 1250 pulses of shockwave therapy on dominant forearm muscles
  Other Names: Dry needle/Acupuncture needle.Shock wave therapy

SUMMARY:
An argument to analyse the Immediate effect of dry needling or extra corporeal shock wave therapy on hand grip strength in normal healthy individuals with a hypothesis of dry needling or shock wave on forearm muscles have influence on the hand grip strength.

DETAILED DESCRIPTION:
After written consent obtained from all the participants randomization and allocation will be done with sealed non transparent envelopes and participants will be assign to two groups Dry needling(DN) and Extra corporeal shock wave therapy (ESWT).Pre and post data of hand grip strength measured with Jamar hand dynamometer.Post data shall be collected precisely after 1 hr of intervention from both groups.

ELIGIBILITY:
Inclusion Criteria:

* No pain on the visual analog scoring scale of 100 mm scale,
* Muscle power of 4+ on oxford manual muscle testing of forearm and wrist extrinsic and intrinsic muscles
* Full range of motion in all dominant upper extremity joints.

Exclusion Criteria:

* History of previous fractures of the dominant upper extremity,
* Teno-synovitis of flexor tendons ,
* Dequervains synovitis,
* Left hand dominance.

Ages: 21 Years to 46 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-11-29 (Actual); Primary Completion 2020-11-29 (Actual); Study Completion 2020-11-29 (Estimated)

PRIMARY OUTCOMES:
Hand Grip Strength | Post 1 hours of Intervention in both groups
  Measurement of Hand Grip Strength with Jamar Dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Rayan M Al-Fadani, BPT, Principal Investigator — Comprehensive rehabilitation centre, Medina Al Munawwarah, Saudi Arabia.; Abdullah M Al-Shenqiti, PhD,PT, Study Director — Taibah University of Medical Rehabilitation Sciences; Tarek M El-Gohary, PhD,PT, Study Chair — Taibah University of Medical Rehabilitation Sciences
Locations (1):
- Comprehensive Rehabilitation Centre, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Results of Hand grip strength pre and post intervention.